CLINICAL TRIAL: NCT03445156
Title: "Boom, Headshot!": Violent First-Person Shooter (FPS) Video Games That Reward Headshots Train Individuals to Aim for the Head When Shooting a Realistic Firearm
Brief Title: Effect of Violent First-Person Shooter (FPS) Video Games on Shooting Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Brad Bushman, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2010B0261
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Gun Shot Wound
Keywords: First-person shooter (FPS); Violent video game; Headshot; Gun; Operant conditioning theory
MeSH Terms: conditions — Wounds, Gunshot | interventions — CDK13 protein, human

STUDY DESIGN:
Intervention Model Description: 2 (controller type) x 3 (video game type) factorial design. Participants used either a regular or gun shaped controller while playing a non-shooting, non-humanoid shooting, or humanoid shooting game.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilot Study (Experimental): After giving their consent, participants completed a survey. Next, they were randomly assigned to play either a violent First-Person-Shooter video game or a nonviolent shooting video game for 20 minutes. Video game play was recorded. A debriefing followed.
  Interventions: Behavioral: Video game; Behavioral: Controller
- Experiment Proper (Experimental): After giving their consent, participants completed a survey. Next, they were randomly assigned to play either a violent First-Person-Shooter video game, a nonviolent shooting video game, or a nonviolent non-shooting video game for 20 minutes. Next, they shot a training pistol at a mannequin 20 feet (6.1 meters) away using 16 Velcro "bullets." A debriefing followed.
  Interventions: Behavioral: Video game; Behavioral: Controller

INTERVENTIONS:
Behavioral: Video game — Participants played either a violent shooting game or nonviolent shooting game in the pilot study, and either either a violent shooting game, nonviolent shooting game, or nonviolent non-shooting game in the experiment proper.
Behavioral: Controller — Participants used either a gun-shaped or regular controller to play the violent and nonviolent shooting video games.

SUMMARY:
The present research tests the effects of violent shooting games on behavior within the game (Pilot Study) and on behavior after the game is turned off (Experiment Proper). The Experiment Proper is an exact replication of a previous study conducted in our lab that was retracted (see citation), but with a larger sample to get more reliable results (N=287 rather than N=151).

DETAILED DESCRIPTION:
Violent shooting games are used to train soldiers and police officers. This research tests whether violent shooting can train people to shoot targets in the head, both during gameplay (Pilot Study) and after the game is turned off (Experiment Proper). Participants in both studies played a violent shooting game with humanoid targets that rewarded headshots, or a nonviolent shooting game that punished shots to bull's-eye targets with faces. Afterward, participants shot at a mannequin with a realistic CO2 gun. We anticipate that participants who play the violent game which rewards headshots to hit the mannequin's head more often than those who play the non-violent game.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Ohio State participant pool

Exclusion Criteria:

* Under age 18

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 327 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-04-25 (Actual); Study Completion 2016-04-25 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
After the manuscript is accepted, data will be uploaded to Figshare.com
Time Frame: Following acceptance of manuscript.
Access Criteria: Open to public domain.

REFERENCES:
- [Background] Whitaker, J. L., & Bushman, B. J. (2014). "Boom, Headshot!": Effect of violent video game play and controller type on firing aim and accuracy. Communication Research, 41(7), 879-891. doi:10.1177/0093650212446622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were college students who completed the study as part of a course requirement.
Pre-assignment Details: After giving their consent, participants completed a survey. Next, they were randomly assigned to play either a violent First-Person-Shooter video game or a nonviolent shooting video game for 20 minutes. Video game play was recorded. A debriefing followed.
Groups:
- Violent Shooter Game: Resident Evil: The Darkside Chronicles, a violent shooter game which rewards players for shooting realistic human targets. Headshots are rewarded.
- Non-violent Shooter Game: Wii Play, a non-violent shooter which punishes players for hitting bull's-eye targets with faces on them and rewards players for shooting other targets (e.g., balloons, clay discs, bull's-eye targets without faces).
- Non-violent Game: Super Mario Galaxy, a non-violent game which rewards players for collecting stars and completing challenging levels in a creative, animated world. Does not involve shooting a weapon.
Period: Pilot Study
Arm/Group | Violent Shooter Game | Non-violent Shooter Game | Non-violent Game
Started | 20 | 20 | 0
Completed | 20 | 20 | 0
Not Completed | 0 | 0 | 0
Period: Experiment Proper
Arm/Group | Violent Shooter Game | Non-violent Shooter Game | Non-violent Game
Started | 113 | 115 | 59
Completed | 113 | 115 | 59
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Undergraduate college students.
Groups:
- Pilot Study: Violent Shooter; Study Proper: Violent Shooter: Resident Evil: The Darkside Chronicles, a violent shooter game which rewards players for shooting realistic human targets. Headshots are rewarded.
- Pilot Study: Non-violent Shooter; Study Proper: Non-violent Shooter: Wii Play, a non-violent shooter which punishes players for hitting bull's-eye targets with faces on them and rewards players for shooting other targets (e.g., balloons, clay discs, bull's-eye targets without faces).
- Study Proper: Non-violent Game: Super Mario Galaxy, a non-violent game which rewards players for collecting stars and completing challenging levels in a creative, animated world. Does not involve shooting a weapon.
- Total: Total of all reporting groups
Arm/Group | Pilot Study: Violent Shooter | Pilot Study: Non-violent Shooter | Study Proper: Violent Shooter | Study Proper: Non-violent Shooter | Study Proper: Non-violent Game | Total
Number analyzed (Participants) | 20 | 20 | 113 | 115 | 59 | 327
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 113 | 115 | 59 | 327
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (1.32) | 19.1 (1.07) | 21.39 (4.27) | 20.70 (2.34) | 20.24 (1.81) | 20.68 (3.06)
Sex: Female, Male [Count of Participants; unit: Participants] — Note: one participant in the study proper did not provide information on their gender. As such, the total is one fewer than the full 327. Population: One participant did not give information on their gender.
  Participants
    number analyzed (Participants) | 20 | 20 | 113 | 115 | 58 | 326
    Female | 10 | 10 | 59 | 61 | 32 | 172
    Male | 10 | 10 | 54 | 54 | 26 | 154
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 113 | 115 | 59 | 327
Gun Attitudes Scale [Mean (Standard Deviation); unit: units on a scale] — 17-item, 5-point Likert scale. Range: 1-5, with higher numbers representing more positive attitudes toward guns. Population: Note: information on attitudes toward guns was not collected in the pilot study
  units on a scale
    number analyzed (Participants) | 0 | 0 | 113 | 115 | 59 | 287
    (all) |  |  | 3.00 (0.70) | 2.96 (0.63) | 2.97 (0.80) | 2.98 (0.69)
Number of guns owned [Mean (Standard Deviation); unit: Number of guns owned] — Participants were asked how many guns (i.e. personal firearms including handguns and long guns) they had owned over the course of their lifetime. Population: Note: information gun ownership was not collected in the pilot study
  Number of guns owned
    number analyzed (Participants) | 0 | 0 | 113 | 115 | 59 | 287
    (all) |  |  | 0.24 (0.88) | 0.23 (0.69) | 0.25 (1.21) | 0.24 (0.89)
Number of times shot gun [Mean (Standard Deviation); unit: number of times shot gun] — Self-report of the number of times each participant had shot a gun (i.e. personal firearm) before. Range: 0 - 550. Population: Information on number of times the participant had shot a gun was not collected in the pilot study.
  number of times shot gun
    number analyzed (Participants) | 0 | 0 | 113 | 115 | 59 | 287
    (all) |  |  | 7.20 (27.55) | 6.15 (20.88) | 14.17 (73.65) | 8.23 (39.88)
Number of violent video games among 3 favorites [Mean (Standard Deviation); unit: Number of games] — Participants were asked to list their three favorite video games. Games rated "T" or "M" by the ESRB were considered violent. Population: Information on favorite games was not collected for the pilot study.
  Number of games
    number analyzed (Participants) | 0 | 0 | 113 | 115 | 59 | 287
    (all) |  |  | 0.72 (0.91) | 0.83 (0.92) | 0.78 (0.91) | 0.78 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Hits to Head and Face
Description: In the Pilot Study, we counted hits to the head and face for targets within the game. In the Experiment Proper, we counted hits to the head and face of the mannequin.
Time Frame: Up to one hour
Measure: Mean (Standard Error); unit: headshots
Groups:
- Pilot Study: Violent Shooter Game; Experiment Proper: Violent Shooter Game: Resident Evil: The Darkside Chronicles, a violent shooter game which rewards players for shooting realistic human targets. Headshots are rewarded.
- Pilot Study: Non-violent Shooter Game; Experiment Proper: Non-violent Shooter Game: Wii Play, a non-violent shooter which punishes players for hitting bull's-eye targets with faces on them and rewards players for shooting other targets (e.g., balloons, clay discs, bull's-eye targets without faces).
- Experiment Proper: Non-violent Game: Super Mario Galaxy, a non-violent game which rewards players for collecting stars and completing challenging levels in a creative, animated world. Does not involve shooting a weapon.
Arm/Group | Pilot Study: Violent Shooter Game | Pilot Study: Non-violent Shooter Game | Experiment Proper: Violent Shooter Game | Experiment Proper: Non-violent Shooter Game | Experiment Proper: Non-violent Game
Number analyzed (Participants) | 20 | 20 | 113 | 115 | 59
headshots | 132.7 (2.68) | 3.88 (37.86) | 5.33 (4.07) | 4.41 (3.77) | 3.86 (3.26)
Statistical Analysis 1: Comparison: Pilot Study: Non-violent Shooter Game; Test type: Other — ANCOVA; p = 0.04, ANCOVA; F(2, 273) = 3.16, p = .044, partial c^2 = .023
Statistical Analysis 2: Comparison: Pilot Study: Violent Shooter Game; Test type: Other — ANCOVA; p = .0001, ANCOVA; F(1, 36) = 44.42

2. Primary Outcome: Other Hits
Description: In the Pilot Study, we counted other hits to targets (i.e. not to a face) within the game. In the Experiment Proper, we counted other hits to the mannequin (i.e., torso instead of the head).
Time Frame: Up to one hour
Measure: Mean (Standard Deviation); unit: shots not at head or face
Arm/Group | Pilot Study: Violent Shooter Game | Pilot Study: Non-violent Shooter Game | Experiment Proper: Violent Shooter Game | Experiment Proper: Non-violent Shooter Game | Experiment Proper: Non-violent Game
Number analyzed (Participants) | 20 | 20 | 113 | 115 | 59
shots not at head or face | 1509.25 (432.41) | 586.10 (145.83) | 6.74 (4.47) | 7.70 (4.39) | 8.03 (5.56)
Statistical Analysis 1: Comparison: Pilot Study: Violent Shooter Game vs Pilot Study: Non-violent Shooter Game; Hypothesis: Participants who played a violent FPS game were expected to have more hits to targets with heads or faces than were participants who played a nonviolent shooting game; Test type: Other — ANCOVA; p < .001, ANCOVA; F(1, 36) = 44.42
Statistical Analysis 2: Comparison: Experiment Proper: Violent Shooter Game vs Experiment Proper: Non-violent Shooter Game vs Experiment Proper: Non-violent Game; Hypothesis: Participants who played a violent FPS game were expected to hit the mannequin's head more often than were participants who played either the nonviolent shooting game or the nonviolent non-shooting game Covariates: participant gender, number of guns owned over their lifetime, attitudes toward guns, and number of times they had fired a gun; Test type: Other — ANCOVA; p = .044, ANCOVA; F(2, 273) = 3.16
Statistical Analysis 3: Comparison: Experiment Proper: Violent Shooter Game vs Experiment Proper: Non-violent Shooter Game vs Experiment Proper: Non-violent Game; Hypothesis: Because the nonviolent shooting game rewards other shots, participants who played a nonviolent shooting game were expected to hit the mannequin's torso more often than were participants who played the nonviolent non-shooting game. Covariates: participant gender, number of guns owned over their lifetime, attitudes toward guns, and number of times they had fired a gun; Test type: Other — ANCOVA; p = 0.17, t-test, 2 sided; t(274) = 2.40
Statistical Analysis 4: Comparison: Experiment Proper: Violent Shooter Game vs Experiment Proper: Non-violent Shooter Game vs Experiment Proper: Non-violent Game; Hypothesis: participants who played a nonviolent shooting game were expected to hit the mannequin's head less often than were participants who played the nonviolent non-shooting game Covariates: participant gender, number of guns owned over their lifetime, attitudes toward guns, and number of times they had fired a gun; Test type: Other — ANCOVA; p = .449, t-test, 2 sided; t(274) = -0.76
Statistical Analysis 5: Comparison: Experiment Proper: Violent Shooter Game vs Experiment Proper: Non-violent Shooter Game vs Experiment Proper: Non-violent Game; Hypothesis: participants who played a nonviolent shooting game were expected to hit the mannequin's torso more often than were participants who played the nonviolent non-shooting game. Covariates: participant gender, number of guns owned over their lifetime, attitudes toward guns, and number of times they had fired a gun; Test type: Other — ANCOVA; p = .645, t-test, 2 sided; t(273) = -0.46
Statistical Analysis 6: Comparison: Experiment Proper: Violent Shooter Game vs Experiment Proper: Non-violent Shooter Game vs Experiment Proper: Non-violent Game; Hypothesis: A positive correlation was expected between the number of violent shooting games participants listed among their three favorite video games and hits to the mannequin's head; Test type: Other — Zero-order correlation; p = .032, Zero-order correlation

ADVERSE EVENTS:
Groups:
- Pilot Study: Violent Shooter: 20 participants assigned to play a violent shooter game
- Pilot Study: Non-violent Shooter: 20 participants assigned to play a non-violent shooter game
- Study Proper: Violent Shooter: 113 participants assigned to play a violent shooter game
- Study Proper: Non-violent Shooter: 115 participants assigned to play a non-violent shooter game
- Study Proper: Non-violent Game: 59 participants assigned to play a non-violent game
Arm/Group | Pilot Study: Violent Shooter | Pilot Study: Non-violent Shooter | Study Proper: Violent Shooter | Study Proper: Non-violent Shooter | Study Proper: Non-violent Game
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/113 | 0/115 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/113 | 0/115 | 0/59
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/113 | 0/115 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes